CLINICAL TRIAL: NCT05298696
Title: Safety and Efficacy of Cilostazol in Prevention of Paclitaxel Induced Peripheral Neuropathy in Breast Cancer Patients
Brief Title: Efficacy of Cilostazol in Prevention of Peripheral Neuropathy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Noha Mansour, Lecturer of Clinical Pharmacy, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2021-395
Record Dates: First submitted 2022-03-17; First posted 2022-03-28 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Peripheral Neuropathy; Breast Cancer
MeSH Terms: conditions — Peripheral Nervous System Diseases; Breast Neoplasms | interventions — Cilostazol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Cilostazol 100 mg twice daily for treatment period
  Interventions: Drug: Cilostazol
- Control (Placebo Comparator): placebo twice daily for treatment period
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cilostazol — Cilostazol 100 mg twice daily
  Arms: Intervention
Drug: Placebo — Placebo twice daily
  Arms: Control

SUMMARY:
There are several mechanisms concerning pathophysiology of paclitaxel induced peripheral neuropathy. One of the main mechanisms is induction of Schwann cell dedifferentiation by paclitaxel. At the preclinical level, cilostazol potently inhibited paclitaxel-induced dedifferentiation of cultured Schwann cells, yet this positive effect have not been clinically investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Breast cancer patients who will receive paclitaxel post-anthracycline therapy.
2. Eastern Cooperative Oncology Group (ECOG) performance status from 0 to 2.
3. Adequate bone marrow function (white blood count ≥4,000/mm3, platelet count≥100,000/mm3), liver function (serum total bilirubin <1.5 mg/dl), renal function (creatinine < 1.5 mg/dl).

Exclusion Criteria:

1. Patients with signs and symptoms of clinical neuropathy at baseline.
2. Patients with diabetes mellitus or alcoholic disease.
3. Patients receiving vitamin/ supplementation drugs that interfere with the study intervention.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Incidence of chemotherapy induced-peripheral neuropathy using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) criteria | 8 weeks post intervention
  Number of patients reported neuropathy from paclitaxel

SECONDARY OUTCOMES:
Severity of chemotherapy induced-peripheral neuropathy | 8 weeks
  Severity of paclitaxel induced peripheral neuropathy using VAS visual analogue scale.
the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity(FACT-GOG-NTX) subscale | 8 weeks
  Measures quality of life related to signs and symptoms of paclitaxel induced peripheral neuropathy
Serum nerve growth factor | 8 weeks
  measuring serum level of nerve growth factor using ELISA KIT
Serum malionaldehyde | 8 weeks
  measuring serum level of maliomaldehyde using spectrophometric kit

OTHER OUTCOMES:
Adverse effects | 8 weeks
  any adverse/ side effect will be evaluated

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Undecided